CLINICAL TRIAL: NCT02856009
Title: Impact of Nutritional Status and Frailty on the Prognosis of Patients Over 75 Years Old Who Suffered a Stroke
Brief Title: Role of Nutrition in Patients Over 75 Years of Age With Stroke
Acronym: INFRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Béjot 2015
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2016-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

ARMS (1):
- patient (Experimental)
  Interventions: Other: completion of a quality of life questionnaire

INTERVENTIONS:
Other: completion of a quality of life questionnaire

SUMMARY:
Stroke in elderly subjects has a more severe clinical presentation (in terms of frequency of aphasia, hemiplegia or consciousness disorders), and a worse functional and vital prognosis. Patients older than 75 years also show excess mortality. One of the hypotheses to explain this situation is the high level of frailty in this population. Many tools to measure the concept of frailty have been developed. One important dimension of these tools is the nutritional status. Indeed, protein-energy malnutrition in the elderly, though a frequent situation, is also a complex phenomenon.

The aim of this study is therefore to analyse the impact of protein-energy malnutrition, as a marker of frailty, on the early prognosis (at 28 days) in the aftermath of stroke in subjects older than 75 years hospitalized in Dijon CHU.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic stroke defined according to WHO criteria (including cerebral infarction and intracerebral haemorrhage) managed at the stroke ICU, Neurology 1, Neurology 2, Internal Medicine 2 or Geriatrics at Dijon CHU during the period from 1st November 2015 to 30th September 2016.
* Patients aged 75 years and older.
* Patients who have provided informed consent to take part in the study.

Exclusion Criteria:

* Patients with meningeal haemorrhage or TIA.
* Patients who refuse to take part in the study.
* Patients with hypo-albuminemia not related to malnutrition: chronic infectious or inflammatory syndrome, nephrotic syndrome, exudative enteropathy, hydration disorders.
* Subjects in custody.
* Patients (or person of trust) who cannot be contacted by telephone during the follow-up.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 177 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Mortality rate | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Dijon, France